CLINICAL TRIAL: NCT06132581
Title: Causal Role of Delta-beta Coupling for Goal-directed Behavior in Anhedonic Depression
Acronym: DBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Justin Riddle, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00004503; 4R00MH126161-03 (NIH)
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder; Anhedonia
Keywords: Transcranial alternating current stimulation; Goal-directed behavior; Cross-frequency coupling
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of three arms of the study: delta-beta tACS, control tACS in theta-gamma, or active sham tACS.
Who Masked: Participant, Investigator
Masking Description: This study is designed to be double-blind. Participants and the researchers are unaware of each participant's assignment until the completion of all data collection. This is accomplished using randomization codes. Furthermore, this study utilizes an active sham stimulation. This means that the active sham condition includes some stimulation, mimicking the skin sensations associated with tACS. In a previously concluded trial, participants in the delta-beta tACS, theta-gamma tACS, and active sham groups responded similarly to the blinding questionnaire, indicating that the active sham stimulation successfully blinded the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Delta-beta tACS (Experimental): The study is investigating the use of transcranial alternating current stimulation (tACS). The stimulation is delivered at 1 milliampere (mA) zero-to-peak amplitude at the target electrodes and 2 mA zero to-peak amplitude at the return electrode. For the experimental arm, the tACS will be delivered using the cross-frequency stimulation waveform delta-beta (3-20Hz).
  Interventions: Device: Delta-beta tACS via the Neurocare Direct Current Stimulator Multi-Channel 4
- Theta-gamma tACS (Active Comparator): This arm serves as an active control where tACS will be delivered using the cross-frequency stimulation waveform theta-gamma (5-50Hz).
  Interventions: Device: Theta-gamma tACS via the Neurocare Direct Current Stimulator Multi-Channel 4
- Active-sham tACS (Sham Comparator): For active sham stimulation, either delta-beta or theta-gamma stimulation is delivered for 15 seconds only at the beginning and end of the stimulation period. This is intended to mimic the skin sensations (e.g., itching, burning, tingling) that are experienced at the onset and offest of stimulation, assisting with blinding the participant's assignment.
  Interventions: Device: Sham tACS via the Neurocare Direct Current Stimulator Multi-Channel 4

INTERVENTIONS:
Device: Delta-beta tACS via the Neurocare Direct Current Stimulator Multi-Channel 4 — Stimulation will be delivered via the Neurocare Direct Current Stimulator Multi-Channel 4, an investigational electrical non-invasive brain stimulation device that is being used for foundational neuroscience and translational research. The electrical waveform for stimulation was designed to mimic delta-beta coupling in the brain.
  Arms: Delta-beta tACS
Device: Theta-gamma tACS via the Neurocare Direct Current Stimulator Multi-Channel 4 — Stimulation will be delivered via the Neurocare Direct Current Stimulator Multi-Channel 4, an investigational electrical non-invasive brain stimulation device that is being used for foundational neuroscience and translational research. The electrical waveform for stimulation was designed to mimic theta-gamma coupling in the brain and is used as an active comparator.
  Arms: Theta-gamma tACS
Device: Sham tACS via the Neurocare Direct Current Stimulator Multi-Channel 4 — Stimulation will be delivered via the Neurocare Direct Current Stimulator Multi-Channel 4, an investigational electrical non-invasive brain stimulation device that is being used for foundational neuroscience and translational research. The electrical waveform is randomly selected to be the theta-gamma or delta-beta waveform, but the stimulation is delivered for only a brief period of time of approximately 30 seconds, which is not sufficient to produce a meaningful dose to the brain. This placebo, or sham, stimulation is designed to mimic the sensation of receiving stimulation.
  Arms: Active-sham tACS

SUMMARY:
Anhedonia, the inability to seek-out and experience pleasure, is a common symptom in depression that predicts treatment-resistance and is sometimes exacerbated by first-line antidepressants. In our previous research, we found that anhedonia decreases goal-directed behavior and its related neural activity. In this study, we will investigate target engagement from five-consecutive days of stimulation for participants that are within a unipolar major depressive episode and also have high symptoms of anhedonia.

DETAILED DESCRIPTION:
The experiment comprises eight sessions total. People that request to be in the experiment will first complete demographic and self-report clinical assessments. People that meet our eligibility criteria will be invited to participate in the study. In the first session, clinical assessment are administered to determine eligibility for the full study. In the second session, participants complete a functional magnetic resonance imaging (MRI) session in which they complete three different reward-based decision-making tasks. After the MRI session, participants are randomized into one of three parallel arms to receive five consecutive days of cross-frequency transcranial alternating current stimulation (CF-tACS) in either delta-beta, control-frequency (theta-gamma), or placebo (sham) CF-tACS. In the third through seventh session, participants receive 40 minutes of CF-tACS while completing goal-setting and action planning worksheets. Before the first session of CF-tACS (the third session overall) and the last session of CF-tACS (the seventh session overall), participants complete brief self-report clinical assessments. On the third and seventh session (the first and fifth day of CF-tACS), the participant will complete the reward-based decision-making tasks prior to stimulation while EEG is recorded. In these two sessions, resting-state EEG is acquired before and after stimulation. The first and fifth session of tACS (third and seventh session overall) will take approximately three hours to complete. The second through fourth session of tACS (fourth through sixth session overall) will take approximately one hour to complete. In the follow-up session, visit 8, (approximately two weeks after the end of the five-days of stimulation), participants return for an in-person session that includes self-report clinical assessments and EEG during the reward-based decision-making tasks.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Able to provide informed consent
* Have normal to corrected vision
* Willing to comply with all study procedures and be available for the duration of the study
* Speak and understand English
* Mild suicide risk as determined by the Hamilton Depression Rating Scale (HAM-D; less than 3 for the suicidality item) and non-existent or mild risk according to the Depression Symptom Index Suicidality Subscale (DSI-SS).
* Patient Health Questionnaire (PHQ-8) greater than or equal to 8 prior to the first session
* Snaith Hamilton Pleasure Scale (SHAPS) greater than 33 at the first session
* A diagnosis of major depressive disorder on the Mini International Neuropsychiatric Interview for the DSM-V (MINI)

Exclusion Criteria:

* ADHD (currently under treatment)
* Neurological disorders and conditions including, but not limited to history of epilepsy; seizures, except childhood febrile seizures; dementia; history of stroke; Parkinson's disease, multiple sclerosis, cerebral aneurysm; brain tumors
* Medical or neurological illness or treatment for a medical disorder that could interfere with study participation. For example, unstable cardiac disease, HIV/AIDS, malignancy, liver or renal impairment
* Prior brain surgery
* Any brain devices/implants including cochlear implants and aneurysm clips, cardiac pacemaker, or any other implanted electronic device
* History of current traumatic brain injury
* Pregnancy (for females)
* Current severe substance use disorder
* Claustrophobia
* Based on the use of MRI, additional exclusion/inclusion criteria are considered. Note that many contraindications for stimulation are common with MRI and thus are not repeated. Participants must not have metal in the body that is ferrous, will be required to remove all jewelry, must not have tattoos on the face or neck, must refrain from wearing metal in clothing (underwire) or active gear (possibility of metallic microparticle technology), must not be a metal worker or have an eye injury involving metal.
* Anything that in the opinion of the investigator would place the participant at increased risk or preclude the participant's full compliance with or completion of the study
* DSM-V diagnosis of present moderate or severe substance use disorder or alcohol use disorder, and past severe substance use disorder or alcohol use disorder, or psychotic disorder within the last 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in coupling strength between prefrontal and posterior cortex | 1 week
  Phase-amplitude coupling strength is calculated between the phase of low-frequency activity in prefrontal electrodes and amplitude of high-frequency in posterior cortex. These signals are extracted from the S-EEfRT during the decision period. Instantaneous phase and amplitude will be calculated by averaging electrodes in the regions, band-filtering to the specified range, and performing the Hilbert transform. Next, a hybrid signal is created using the high-frequency amplitude and low-frequency phase. Coupling strength is the magnitude of the average of this signal over time. Finally, coupling strength is normalized using a z-transformation with respect to a null distribution generated by randomly time-shifting the high-frequency time-series.

SECONDARY OUTCOMES:
Change in Symptoms of anhedonia | 4 weeks
  Anhedonia is measured using the Snaith Hamilton Pleasure Rating Scale (SHAPS) which ranges from 14 to 56 where a larger value reflects greater symptoms of anhedonia.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with FSU.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from 9 to 36 months following publication
Access Criteria: Deidentified individual data that supports the results will be shared provided the investigator who proposes to use the data has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with FSU.